CLINICAL TRIAL: NCT00218023
Title: Screening Medications for Cocaine Cessation and Relapse Prevention
Brief Title: Medications for Stopping Cocaine Dependence and Preventing Relapse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Joy Schmitz, Professor - Psy, Behavioral Science, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-09262-7; P50DA009262-07 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Cocaine Abuse; Cocaine-Related Disorders
Keywords: cocaine; cocaine addiction; cocaine abuse; relapse prevention
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Modafinil; carbidopa, levodopa drug combination; Naltrexone; Motivational Interviewing; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Modafinil plus MI, CM, and CBT (Experimental): The modafinil dose began at 200 mg (day 1) and increased to the fixed dose of 200 mg twice daily (day 2) during the 12 weeks of Phase II.
  The motivational interviewing (MI) intervention consisted of two 1-h individual therapy sessions on the first and eighth day of Phase I.
  Contingency management (CM) is a voucher-based intervention. Subjects earned vouchers for cocaine abstinence (during Phase I) and medication compliance (during Phase II).
  Subjects received weekly, 1-h, individual Cognitive-Behavioral Therapy (CBT) sessions during Phase II.
  Interventions: Drug: Modafinil; Behavioral: Motivational Interviewing (MI); Behavioral: Contingency management (CM); Behavioral: Cognitive-Behavioral Therapy (CBT)
- Levodopa/Carbidopa plus MI, CM, and CBT (Experimental): Levodopa-carbidopa, in the sustained-release formulation (Sinemet CR), began at a dose of levodopa/carbidopa 400/100 mg (day 1) and increased to the fixed dose of 400/100 mg twice daily (day 2) during the 12 weeks of Phase II.
  The motivational interviewing (MI) intervention consisted of two 1-h individual therapy sessions on the first and eighth day of Phase I.
  Contingency management (CM) is a voucher-based intervention. Subjects earned vouchers for cocaine abstinence (during Phase I) and medication compliance (during Phase II).
  Subjects received weekly, 1-h, individual Cognitive-Behavioral Therapy (CBT) sessions during Phase II.
  Interventions: Drug: Levodopa/Carbidopa; Behavioral: Motivational Interviewing (MI); Behavioral: Contingency management (CM); Behavioral: Cognitive-Behavioral Therapy (CBT)
- Naltrexone HCl plus MI, CM, and CBT (Experimental): Naltrexone hydrochloride (HCl) doses began at 25 mg (day 1) and increased to the fixed dose of 25 mg twice daily (day 2) during the 12 weeks of Phase II.
  The motivational interviewing (MI) intervention consisted of two 1-h individual therapy sessions on the first and eighth day of Phase I.
  Contingency management (CM) is a voucher-based intervention. Subjects earned vouchers for cocaine abstinence (during Phase I) and medication compliance (during Phase II).
  Subjects received weekly, 1-h, individual Cognitive-Behavioral Therapy (CBT) sessions during Phase II.
  Interventions: Drug: Naltrexone HCl; Behavioral: Motivational Interviewing (MI); Behavioral: Contingency management (CM); Behavioral: Cognitive-Behavioral Therapy (CBT)
- Placebo plus MI, CM, and CBT (Placebo Comparator): Placebo capsules were identical in appearance to active drug capsules, and each contained 50 mg riboflavin for subsequent evaluation of medication compliance.
  The motivational interviewing (MI) intervention consisted of two 1-h individual therapy sessions on the first and eighth day of Phase I.
  Contingency management (CM) is a voucher-based intervention. Subjects earned vouchers for cocaine abstinence (during Phase I) and medication compliance (during Phase II).
  Subjects received weekly, 1-h, individual Cognitive-Behavioral Therapy (CBT) sessions during Phase II.
  Interventions: Drug: Placebo; Behavioral: Motivational Interviewing (MI); Behavioral: Contingency management (CM); Behavioral: Cognitive-Behavioral Therapy (CBT)

INTERVENTIONS:
Drug: Modafinil — The modafinil dose began at 200 mg (day 1) and increased to the fixed dose of 200 mg twice daily (day 2) during the 12 weeks of Phase I.
  Other Names: Provigil
  Arms: Modafinil plus MI, CM, and CBT
Drug: Levodopa/Carbidopa — Levodopa-carbidopa, in the sustained-release formulation (Sinemet CR), began at a dose of levodopa/carbidopa 400/100 mg (day 1) and increased to the fixed dose of 400/100 mg twice daily (day 2) during the 12 weeks of Phase I.
  Other Names: Simemet CR
  Arms: Levodopa/Carbidopa plus MI, CM, and CBT
Drug: Naltrexone HCl — Naltrexone hydrochloride (HCl) doses began at 25 mg (day 1) and increased to the fixed dose of 25 mg twice daily (day 2) during the 12 weeks of Phase I.
  Other Names: Naltrexon hydrochloride
  Arms: Naltrexone HCl plus MI, CM, and CBT
Drug: Placebo — Placebo capsules were identical in appearance to active drug capsules, and each contained 50 mg riboflavin for subsequent evaluation of medication compliance.
  Arms: Placebo plus MI, CM, and CBT
Behavioral: Motivational Interviewing (MI) — The primary goal of motivational interviewing (MI) was to assist patients in achieving initial abstinence by increasing motivation and commitment to change. The MI intervention consisted of two 1-h individual therapy sessions on the first and eighth day of Phase I. The client-centered, MI-style sessions focused on building motivation for change, exploring ambivalence, obtaining a commitment to change, making a plan for abstinence (Session 1), providing personalized feedback, reassessing commitment for change, and reevaluating the change plan (Session 2). Masters-level therapists were trained and supervised by the therapy supervisor (ALS), an expert in motivation-based therapies.
Behavioral: Contingency management (CM) — Contingency management (CM) is a voucher-based intervention. Subjects earned vouchers for cocaine abstinence (during phase I) and medication compliance (during phase II).
Behavioral: Cognitive-Behavioral Therapy (CBT) — Subjects received weekly, 1-h, individual Cognitive-Behavioral Therapy (CBT) sessions during Phase II. This therapy component focused on coping-skills training for resisting cocaine use in high-risk situations, based on relapse-prevention theory and manual-guided techniques. Therapy sessions were conducted by master's-level licensed professional counselors supervised by a licensed clinical psychologist, who monitored manual adherence and competency.

SUMMARY:
Cocaine dependence is a major public health problem; an effective primary treatment for cocaine dependent individuals has yet to be found. The purpose of this study is to identify subpopulations and baseline conditions that are most responsive to treatment for cocaine dependent individuals.

DETAILED DESCRIPTION:
Cocaine is a strong central nervous system stimulant that is widely abused throughout the United Sates. Due to its widespread use, it is important to develop an effective treatment for cocaine dependence. Motivational Interviewing (MI) is often effective when combined with drug treatment. Baseline condition (e.g., abstinence status) and population type (e.g., ethnicity and gender) often affect how an individual responds to treatment for drug dependence. The purpose of this study is to determine the influence of baseline status and population type on treatment response in cocaine dependent individuals. In addition, this study will examine how various cocaine abuse medications target different neuronal systems, withdrawal symptoms, and relapse to drug use.

This study will take place in two phases. Phase I will last 4 weeks; participants will receive MI and undergo contingency-based urine tests in order to achieve the desired baseline condition. Phase II will last 12 weeks. Participants in Phase II will be randomly assigned to receive one of four treatments: 1) 50 mg naltrexone, 2) 800/200 mg levodopa/carbidopa, 3) 400 mg modafinil, or 4) placebo. During Phase II, all participants will receive psychotherapy and contingency management. Participants will complete urine drug screening tests 3 times each week. Follow-up study visits will occur between 3 and 6 months following Week 12, and will include objective and self-reported drug use.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for current cocaine dependence

Exclusion Criteria:

* Meet diagnostic criteria for other serious psychiatric symptoms and/or disorders that would interfere with participation in the treatment study (e.g., psychosis; mania; suicidal/ homicidal ideation) including other forms of drug dependence, nicotine and cannabis excepted.
* Medical conditions contraindicating naltrexone therapy (e.g., past history of opioid use in the 30 days prior to study entry or significant hepatocellular injury)
* Medical conditions contraindicating modafinil therapy (e.g., hypertension, seizures, arrhythmia, or coronary artery disease)
* Medical conditions contraindicating levodopa/carbidopa therapy (e.g., severe pulmonary/cardiovascular disease, narrow angle glaucoma, melanoma, history of peptic ulcer, or renal function impairment)
* Requires certain medications
* Current or recent treatment for substance use or other psychiatric condition
* On parole or probation that requires reports of drug use to officers of the court
* Pending incarceration
* Pregnant or breastfeeding
* Unable to read, write, or speak English
* Plans to leave the study area within 3 months of study entry

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2006-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joy M Schmitz, PhD, Principal Investigator — University of Texas
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Result] Schmitz JM, Green CE, Stotts AL, Lindsay JA, Rathnayaka NS, Grabowski J, Moeller FG. A two-phased screening paradigm for evaluating candidate medications for cocaine cessation or relapse prevention: modafinil, levodopa-carbidopa, naltrexone. Drug Alcohol Depend. 2014 Mar 1;136:100-7. doi: 10.1016/j.drugalcdep.2013.12.015. Epub 2014 Jan 3. PMID 24424425

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 101 subjects were enrolled and began phase 1 (in phase 1, all enrolled subjects received the same intervention, motivational interviewing, which is described in the Interventions section). 81 completed phase 1, and 81 started phase 2, as described in the Period below. Subjects were assigned to the 4 arms at phase 2.
Period: Overall Study
Arm/Group | Modafinil Plus MI, CM, and CBT | Levodopa/Carbidopa Plus MI, CM, and CBT | Naltrexone HCl Plus MI, CM, and CBT | Placebo Plus MI, CM, and CBT
Started (Number that started phase 2, the phase in which subjects were assigned to the 4 arms.) | 22 | 25 | 16 | 18
Received Drug or Placebo in Phase II | 18 | 24 | 15 | 18
Completed | 9 | 10 | 6 | 11
Not Completed | 13 | 15 | 10 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modafinil Plus MI, CM, and CBT | Levodopa/Carbidopa Plus MI, CM, and CBT | Naltrexone HCl Plus MI, CM, and CBT | Placebo Plus MI, CM, and CBT | Total
Number analyzed (Participants) | 22 | 25 | 16 | 18 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.64 (5.71) | 40.66 (8.6) | 42.08 (9.89) | 42.29 (10.5) | 42.16 (8.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 4 | 1 | 14
  Male | 19 | 19 | 12 | 17 | 67
Region of Enrollment [Number; unit: participants]
  United States | 22 | 25 | 16 | 18 | 81

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage of Cocaine-positive Urines Over Course of 12 Week Treatment in Subgroup Achieving Abstinence at Baseline
Description: Cocaine use was determined by assessing for the presence of benzoylecgonine in urine.
Time Frame: 3 times per week (Monday, Wednesday, and Friday) for 12 weeks
Measure: Mean (Standard Error); unit: Mean % of cocaine-positive urines
Arm/Group | Modafinil Plus MI, CM, and CBT | Levodopa/Carbidopa Plus MI, CM, and CBT | Naltrexone HCl Plus MI, CM, and CBT | Placebo Plus MI, CM, and CBT
Number analyzed (Participants) | 8 | 8 | 9 | 10
Mean % of cocaine-positive urines | 31 (0.238) | 28 (0.20) | 47 (0.261) | 35 (0.186)

2. Primary Outcome: Mean Percentage of Cocaine-positive Urines Over Course of 12 Week Treatment in Subgroup NOT Achieving Abstinence at Baseline
Description: Cocaine use was determined by assessing for the presence of benzoylecgonine in urine.
Time Frame: 3 times per week (Monday, Wednesday, and Friday) for 12 weeks
Measure: Mean (Standard Error); unit: Mean % of cocaine-positive urines
Arm/Group | Modafinil Plus MI, CM, and CBT | Levodopa/Carbidopa Plus MI, CM, and CBT | Naltrexone HCl Plus MI, CM, and CBT | Placebo Plus MI, CM, and CBT
Number analyzed (Participants) | 14 | 17 | 7 | 8
Mean % of cocaine-positive urines | 88 (0.029) | 49 (0.254) | 62 (0.219) | 91 (0.016)

ADVERSE EVENTS:
Time Frame: The 12 weeks during which the drugs were administered (i.e., Phase II).
Arm/Group | Modafinil Plus MI, CM, and CBT | Levodopa/Carbidopa Plus MI, CM, and CBT | Naltrexone HCl Plus MI, CM, and CBT | Placebo Plus MI, CM, and CBT
Serious Adverse Events (participants affected / at risk) | 1/22 | 4/25 | 1/16 | 1/18
Other Adverse Events (participants affected / at risk) | 0/22 | 0/25 | 0/16 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modafinil Plus MI, CM, and CBT (N=22) | Levodopa/Carbidopa Plus MI, CM, and CBT (N=25) | Naltrexone HCl Plus MI, CM, and CBT (N=16) | Placebo Plus MI, CM, and CBT (N=18)
eye injury (torn conjunctiva) (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
arrhythmia symptoms (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
suicidal tendencies (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
routine liver-function tests showed an increase from baseline in hepatic enzyme values (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
work-related traumatic injury to finger that required surgical repair (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The sample size was small; however, the main aim of the study was achieved (i.e., to evaluate the feasibility of using a two-phase abstinence induction paradigm to screen candidate medications for cocaine treatment).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes